CLINICAL TRIAL: NCT01843621
Title: A Phase I/II, Open, Five-year, Clinical Follow-up Study of Thai Children Who Participated in Dengue-003 ("A Phase I/II Trial of a Tetravalent Live Attenuated DEN Vaccine in Flavivirus Antibody Naive Children") With Evaluation of a Booster Dose Given One Year After Primary DEN Vaccination Series
Brief Title: A Phase I/II Trial of a Tetravalent Live Attenuated DEN Vaccine in Flavivirus Antibody Naive Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-13227; GSK 103795 (Other: GSK); WRAIR 1159 (Other: WRAIR); NCT00318916 (obsolete NCT alias)
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-05

CONDITIONS: Dengue
Keywords: Dengue, Vaccine, Thailand
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Total vaccinated (Experimental): The total vaccinated cohort included all enrolled subjects who received the DEN vaccine F17 for whom data were available. These subjects were Thai children previously enrolled and vaccinated in study Dengue-003
  Interventions: Biological: DEN vaccine F17

INTERVENTIONS:
Biological: DEN vaccine F17 — The dengue booster vaccine was administered subcutaneously in the non-dominant arm (deltoid). The tetravalent, live attenuated DEN F17 vaccine was administered in this study. This pre-transfection formulation contained dengue virus types 1, 2, 3 and 4 (DEN-1, -2, -3 and -4).
  Other Names: Live attenuated tetravalent dengue (DEN) vaccine

SUMMARY:
One year follow-up on immunogenicity and safety of a booster dose of DEN vaccine administered approx. 1 year following the second dose

DETAILED DESCRIPTION:
The purpose of this study is to find out more about the two doses of dengue vaccine, over a five year period, that the children received in the Dengue-003 study and to study a third dose of dengue that will be given to the children

* Do children still have dengue antibodies intended to provide protection against dengue infection one year after the two doses of vaccine given in study Dengue-003?
* Were there any major medical problems that appeared as dengue-like symptoms during the one year after vaccinations?
* Will a third dose of dengue help to further stimulate the part of the immune system intended to help protect against dengue infection?
* Is a third dose as safe as the first two doses?
* Are the local reactions to a third dose of the vaccine similar to what your child experienced after the first two doses?

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received two doses of DEN vaccine in the Dengue-003 study
* Subjects whos parents signed an informed consent form were eligible for participation in the five year follow-up study

Exclusion Criteria:

* None

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2005-02; Primary Completion 2005-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriluck Simasathien, M.D., Principal Investigator — Department of Pediatrics, Phramongkutklao Hospital, Bangkok, Thailand; Robert Gibbons, M.D., Principal Investigator — Armed Forces Research Institute of Medical Sciences (AFRIMS), Bangkok, Thailand
Locations (1):
- Department of Pediatrics, Phramongkutklao Hospital, Phayathai, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
GSK

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven Thai children from the Dengue-03 study will be invited to participate
Period: Overall Study
Arm/Group | Total Vaccinated
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (0.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  Thailand | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seropositivity Rates for Antibodies to DEN-1 - DEN-4 (ATP Cohort for Immunogenicity)
Description: Neutralizing antibodies as measured by plaque reduction neutralization test (seropositivity rates to each dengue virus serotype at Prebooster Year 1, 30 Days Post Booster, Year 2, and Year 3 time points.
Time Frame: Prebooster Year 1, 30 Days Post Booster, Year 2, and Year 3
Population: Immunogenicity data for one subject was not included in the ATP analysis due to an asymptomatic, sub-clinical, wild-type DEN-2 virus infection prior to DEN vaccine dose 1
Measure: Mean (95% Confidence Interval); unit: % of subjects
Groups:
- > 10 ED50: Seropositivity rates (% of subjects)
Arm/Group | > 10 ED50
Number analyzed (Participants) | 6
% of subjects
  N lg to DEN-1: Prebooster Year 1 | 16.7 [0.4 to 64.1]
  N lg to DEN-1: 30 Days Post Booster | 83.3 [35.9 to 99.6]
  N lg to DEN-1: Year 2 | 16.7 [0.4 to 64.1]
  N lg to DEN-1: Year 3 | 66.7 [22.3 to 95.7]
  N lg to DEN-2: Prebooster Year 1 | 50.0 [11.8 to 88.2]
  N lg to DEN-2: 30 Days Post Booster | 100 [54.1 to 100]
  N lg to DEN-2: Year 2 | 66.7 [22.3 to 95.7]
  N lg to DEN-2: Year 3 | 83.3 [35.9 to 99.6]
  N lg to DEN-3: Prebooster Year 1 | 33.3 [4.3 to 77.7]
  N lg to DEN-3: 30 Days Post Booster | 100 [54.1 to 100]
  N lg to DEN-3: Year 2 | 33.3 [4.3 to 77.7]
  N lg to DEN-3: Year 3 | 50.0 [11.8 to 88.2]
  N lg to DEN-4: Prebooster Year 1 | 50.0 [11.8 to 88.2]
  N lg to DEN-4: 30 days Post Booster | 100 [54.1 to 100]
  N lg to DEN-4: Year 2 | 50.0 [11.8 to 88.2]
  N lg to DEN-4: Year 3 | 100 [54.1 to 100]

2. Primary Outcome: Geometric Mean Titers (GMTs) on All Subjects for Antibodies to DEN-1 - DEN-4 (ATP Cohort for Immunogenicity)
Description: Neutralizing antibodies as measured by plaque reduction neutralization test (geometric mean titers [GMTs]) to each dengue virus serotype at Prebooster Year 1, 30 Days Post Booster, Year 2, and Year 3 time points.
Time Frame: Prebooster Year 1, 30 Days Post Booster, Year 2, and Year 3
Measure: Mean (95% Confidence Interval); unit: GMTs
Groups:
- Geometric Mean Titer (GMT): Geometric mean antibody titer value
Arm/Group | Geometric Mean Titer (GMT)
Number analyzed (Participants) | 6
GMTs
  N lg to DEN-1: Pre-booster Year 1 | 6.0 [3.8 to 9.6]
  N lg to DEN-1: 30 Days Post-booster | 28.2 [6.6 to 121.3]
  N lg to DEN-1: Year 2 | 6.8 [3.1 to 15.1]
  N lg to DEN-1: Year 3 | 18.0 [5.2 to 63.0]
  N lg to DEN-2: Pre-booster Year 1 | 16.8 [3.4 to 82.5]
  N lg to DEN-2: 30 Day Post-booster | 94.4 [24.0 to 370.3]
  N lg to DEN-2: Year 2 | 20.8 [4.6 to 92.9]
  N lg to DEN-2: Year 3 | 36.3 [7.0 to 186.8]
  N lg to DEN-3: Pre-booster Year 1 | 12.8 [2.1 to 77.5]
  N lg to DEN-3: 30 Days post-booster | 67.2 [9.3 to 487.2]
  N lg to DEN-3: Year 2 | 9.4 [2.8 to 31.7]
  N lg to DEN-3: Year 3 | 12.9 [4.1 to 41.3]
  N lg to DEN-4: Pre-booster Year 1 | 27.0 [3.6 to 200.7]
  N lg to DEN-4: 30 Days Post-booster | 112.0 [26.5 to 473.1]
  N lg to DEN-4: Year 2 | 25.4 [3.5 to 182.1]
  N lg to DEN-4: Year 3 | 70.4 [23.9 to 207.4]

3. Secondary Outcome: Solicited Local Adverse Events (AEs) Within 21 Day Follow-up
Description: Incidence of solicited local symptoms reported during the 21-day post-vaccination (total vaccination cohort).
Time Frame: 21 days
Population: Incidence of solicited local symptoms reported during the 21-day post-vaccination (total vaccination cohort).
Measure: Number; unit: Adverse events
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Adverse events
  Pain: All | 3
  Pain: Grade 3 | 0
  Redness: All | 3
  Redness: Grade 3 | 0
  Swelling: All | 4
  Swelling: Grade 3 | 1

4. Secondary Outcome: Unsolicited Adverse Events (AEs) Within 31 Days Post Vaccination
Description: Percentage of subjects reporting unsolicited AEs within 31 days (Day 0-30) after the DEN vaccine dose (total vaccinated cohort)
Time Frame: 31 days
Population: Percentage of subjects reporting unsolicited AEs within 31 days (Day 0-30) after the DEN vaccine dose (total vaccinated cohort)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Percentage of subjects
  At Least One Symptom | 85.7 [42.1 to 99.6]
  Infections and Infestations | 14.3 [0.4 to 57.9]
  Injury, Poisoning and Procedural Complications | 14.3 [0.4 to 57.9]
  Nervous System Disorders | 42.9 [9.9 to 81.6]
  Renal and Urinary Disorders | 14.3 [0.4 to 57.9]
  Respiratory, Thoracic and Mediastinal Disorders | 28.6 [3.7 to 71.0]

5. Secondary Outcome: Serious Adverse Events (SAE) Within 31 Days Post Vaccination
Description: Occurrence of SAEs within 31 days (Day 0-30) after vaccination
Time Frame: 31 days
Population: Occurrence of SAEs within 31 days (Day 0-30) after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Participants | 0

6. Secondary Outcome: Abnormal Findings Reported During Physical Exam 31-Days Post Vaccination
Description: Incidence of dengue physical examination findings reported during the 31-day post-vaccination period (total vaccinated cohort)
Time Frame: 31 days
Population: Incidence of dengue physical examination findings reported during the 31-day post-vaccination period (total vaccinated cohort)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Percentage of subjects | 42.9 [9.9 to 86.6]

7. Secondary Outcome: Monovalent, Bivalent, Trivalent and Tetravalent Response for Neutralizing Antibodies 30 Days Post Booster
Description: Monovalent, Bivalent, Trivalent and Tetravalent response for DEN neut. antibodies 30 days post booster dose vaccine (ATP cohort for immunogenicity)
Time Frame: Prebooster year 1, 30 Days Post Booster, Year 2, Year 3
Population: Monovalent, Bivalent, Trivalent and Tetravalent response for DEN neut. antibodies 30 days post booster dose vaccine (ATP cohort for immunogenicity). Immunogenicity data for one subject was not included in the ATP analysis due to an asymptomatic, sub-clinical, wild-type DEN-2 virus infection prior to DEN vaccine dose 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 6
percentage of subjects
  Pre-Booster Year 1: Monovalent | 16.67 [0.42 to 64.12]
  Pre-Booster Year 1: Bivalent | 33.33 [4.33 to 77.72]
  Pre-Booster Year 1: Trivalent | 0.00 [0.00 to 45.93]
  Pre-Booster Year 1: Tetravalent | 16.67 [0.42 to 64.12]
  30 Days Post Booster: Monovalent | 0.00 [0.00 to 45.93]
  30 Days Post Booster: Bivalent | 0.00 [0.00 to 45.93]
  30 Days post Booster: Trivalent | 16.67 [0.42 to 64.12]
  30 Days Post Booster: Tetravalent | 83.33 [35.88 to 99.58]
  Year 2: Monovalent | 33.33 [4.33 to 77.72]
  Year 2: Bivalent | 33.33 [4.33 to 77.72]
  Year 2: Trivalent | 0.00 [0.00 to 45.93]
  Year 2: Tetravalent | 16.67 [0.42 to 64.12]
  Year 3: Monovalent | 0.00 [0.00 to 45.93]
  Year 3: Bivalent | 33.33 [4.33 to 77.72]
  Year 3: Trivalent | 33.33 [4.33 to 77.72]
  Year 3: Tetravalent | 33.33 [4.33 to 77.72]

8. Secondary Outcome: Presence of Dengue Viremia 10 Days After the Dengue Vaccine Dose
Description: Nested Polymerase Chain Reaction (PCR) for DEN was conducted on day 10 after DEN booster vaccination to evaluate the presence of Dengue viremia 10 days after vaccination
Time Frame: 10 days
Population: Nested PCR for DEN was conducted on day 10 after DEN booster vaccination to evaluate the presence of Dengue viremia 10 days after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Total Vaccinated
Number analyzed (Participants) | 7
Participants | 1

9. Secondary Outcome: Flavivirus Infection in Terms of Dengue Immunoglobulin M and Immunoglobulin G Per Subject (ATP Cohort for Immunogenicity)
Description: The ratio of DEN Immunoglobulin type M and G (IgM:IgG) measured at the time of booster vaccination and 30 days following was used to assess intercurrent flavivirus infection. Flavivirus infection in terms of dengue IgM and IgG and Japanese encephalitis virus (JEV) IgM and IgG is summarized.
  Flavivirus immunity= ratio IgM on IgG <1.8 with either IgM or IgM >1:40
  If the antibody response is detectable by isotype capture enzyme immunoassay (either the IgM or IgG component ≥40 U), its anamnestic character can be inferred from detection of a DEN IgM to IgG ratio of <1.8.
Time Frame: 1 year, 30 Days Post Booster, 2 years
Measure: Number; unit: Flavivirus immunity ratio
Groups:
- Ratio IgM and IgG: Ratio of Dengue (DEN) IgM and IgG and Japanese encephalitis virus (JEV) IgM and IgG (ATP cohort for immunogenicity)
Arm/Group | Ratio IgM and IgG
Number analyzed (Participants) | 6
Flavivirus immunity ratio
  DEN Subject 2: 1 Year Ratio | 0
  DEN Subject 2: 30 Days Post Booster Ratio | 0.3
  DEN Subject 2: Year 2 Ratio | 0
  JEV Subject 2: Year 1 Ratio | 0
  JEV Subject 2: 30 Days Post Booster Ratio | 0.4
  JEV Subject 2: Year 2 Ratio | 0
  DEN Subject 3: Year 1 Ratio | 0
  DEN Subject 3: 30 Days Post Booster Ratio | 0
  DEN Subject 3: Year 2 Ratio | 0
  JEV Subject 3: Year 1 Ratio | 0
  JEV Subject 3: 30 Days Post Booster Ratio | 0
  JEV Subject 3: Year 2 Ratio | 0
  DEN Subject 4: Year 1 Ratio | 0
  DEN Subject 4: 30 Days Post Booster Ratio | 0
  DEN Subject 4: Year 2 Ratio | 0
  JEV Subject 4: Year 1 Ratio | 0
  JEV Subject 4: Year 2 Ratio | 0
  DEN Subject 5: Year 1 Ratio | 0
  DEN Subject 5: 30 Days Post Booster Ratio | 0
  DEN Subject 5: Year 2 Ratio | 0
  JEV Subject 5: Year 1 Ratio | 0
  JEV Subject 5: 30 Days Post Booster Ratio | 0
  JEV Subject 5: Year 2 Ratio | 0
  DEN Subject 6: Year 1 Ratio | 0
  DEN Subject 6: 30 Days Post Booster Ratio | 0
  DEN Subject 6: Year 2 Ratio | 0
  JEV Subject 6: Year 1 Ratio | 0
  JEV Subject 6: 30 Days Post Booster Ratio | 0
  JEV Subject 6: Year 2 Ratio | 0
  DEN Subject 7: Year 1 Ratio | 0
  DEN Subject 7: 30 Days Post Booster Ratio | 0
  DEN Subject 7: Year 2 Ratio | 0
  JEV Subject 7: Year 1 Ratio | 0
  JEV Subject 7: 30 Days Post Ratio | 0
  JEV Subject 7: Year 2 Ratio | 0

10. Secondary Outcome: Subject Biochemistry and Hematology Parameters Monitored for Alert Levels
Description: Clinical safety laboratory test were monitored for alert levels. Tests were performed by Laser scattering using Cell Dyn 3500 and Serum chemistry conducted by Kinetic method using Hitachi 717.
  Normal Ranges:
  Alanine Aminotransferases (ALT): LNL=0 and UNL=30 Aspartate Aminotransferases (AST): LNL=0 and UNL=40 Platelet (PLA): LNL=150000 and UNL=350000 Hematocrit (HC): LNL=35 and UNL=45 Neutrophil (NEU): LNL=1500 and UNL=8000
Time Frame: Year 1 (day 0); Year 1 (day 30); Year 2
Population: Tests were performed by Laser scattering using Cell Dyn 3500 and Serum chemistry conducted by Kinetic method using Hitachi 717. Tests included ALT, AST, PLA, HC, and NEU levels.
Measure: Number; unit: U/L
Groups:
- ALT Level: Normal Range = 0-30
- AST Level: Normal Range = 0-40
- PLA Level: Normal Range = 150000-350000
- HC Level: Normal Range = 35-45
- NEU Level: Normal Range = 1500-8000
Arm/Group | ALT Level | AST Level | PLA Level | HC Level | NEU Level
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
U/L
  Subject 1: Year 1, Day 0 | 15 | 28 | 494000 | 37 | 2820
  Subject 1: Year 1, Day 10 | 15 | 34 | 369000 | 37.1 | 3020
  Subject 1: Year 1, Day 30 | 12 | 32 | 411000 | 39.3 | 3000
  Subject 1: Year 2 | 12 | 23 | 502000 | 38.9 | 4790
  Subject 2: Year 1, Day 0 | 10 | 29 | 293000 | 36.1 | 3210
  Subject 2: Year 1, Day 10 | 13 | 30 | 248000 | 36.9 | 2770
  Subject 2: Year 1, Day 30 | 12 | 31 | 296000 | 35.9 | 3070
  Subject 2: Year 2 | 11 | 28 | 323000 | 38.4 | 2400
  Subject 3: Year 1, Day 0 | 51 | 28 | 270000 | 39.3 | 2580
  Subject 3: Year 1, Day 10 | 68 | 44 | 272000 | 41.8 | 3750
  Subject 3: Year 1, Day 30 | 68 | 36 | 303000 | 42.3 | 4380
  Subject 3: Year 2 | 46 | 33 | 306000 | 40.4 | 5170
  Subject 4: Year 1, Day 0 | 11 | 24 | 280000 | 38.8 | 3320
  Subject 4: Year 1, Day 10 | 12 | 23 | 253000 | 39.9 | 3460
  Subject 4: Year 1, Day 30 | 13 | 34 | 297000 | 41.8 | 3320
  Subject 4: Year 2 | 16 | 34 | 231000 | 43.1 | 3900
  Subject 5: Year 1, Day 0 | 49 | 45 | 403000 | 39 | 3950
  Subject 5: Year 1, Day 10 | 28 | 36 | 415000 | 40.2 | 4580
  Subject 5: Year 1, Day 30 | 41 | 49 | 329000 | 38.8 | 2970
  Subject 5: Year 2 | 26 | 29 | 346000 | 36.6 | 5920
  Subject 6: Year 1, Day 0 | 10 | 27 | 440000 | 36.6 | 3020
  Subject 6, Year 1, Day 10 | 13 | 28 | 434000 | 38 | 3390
  Subject 6, Year 1, Day 30 | 12 | 28 | 417000 | 35.4 | 2690
  Subject 6, Year 2 | 16 | 35 | 461000 | 39.7 | 3840
  Subject 7: Year 1, Day 0 | 11 | 27 | 244000 | 38.6 | 3460
  Subject 7: Year 1, Day 10 | 12 | 26 | 238000 | 37.1 | 3050
  Subject 7: Year 1, Day 30 | 10 | 29 | 270000 | 38.4 | 2940
  Subject 7, Year 2 | 13 | 27 | 311000 | 41.4 | 4240

ADVERSE EVENTS:
Time Frame: 21 days post vaccination period following each dose
Arm/Group | Total Vaccinated
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Vaccinated (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — < 2 days
Abdominial Pain (Gastrointestinal disorders) | 0 (0) — > 2 days
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) — < 2 days
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — > 2 days
Fatigue (General disorders) | 4 (4) — < 2 days
Fatigue (General disorders) | 0 (0) — > 2 days
Fever (Axillary) (General disorders) | 1 (1) — < 2 days
Fever (Axillary) (General disorders) | 0 (0) — > 2 days
Headache (Nervous system disorders) | 1 (1) — < 2 days
Headache (Nervous system disorders) | 1 (1) — > 2 days
Muscle aches (Musculoskeletal and connective tissue disorders) | 3 (3) — < 2 days
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) — > 2 days
Nausea (Gastrointestinal disorders) | 0 (0) — < 2 days
Nausea (Gastrointestinal disorders) | 0 (0) — > 2 days
Pain behind eyes (Eye disorders) | 1 (1) — < 2 days
Pain behind eyes (Eye disorders) | 1 (1) — > 2 days
Photophobia (Eye disorders) | 1 (1) — < 2 days
Photophobia (Eye disorders) | 1 (1) — > 2 days
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — < 2 days
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) — > 2 days
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — < 2 days
Rash (Skin and subcutaneous tissue disorders) | 0 (0) — > 2 days
Vomiting (Gastrointestinal disorders) | 0 (0) — < 2 days
Vomiting (Gastrointestinal disorders) | 0 (0) — > 2 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No